CLINICAL TRIAL: NCT04469673
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Efficacy, as Well as Immunogenecity, Pharmacokineticks and Pharmacodynamics of Multiple Doses of JS002 on Stable Statin Therapy in Patients With Hyperlipidemia.
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of Multiple Doses of JS002 in Patients With Hyperlipidemia..
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS002-002
Record Dates: First submitted 2020-07-06; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Hyperlipemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS002 (Experimental): Participants received one of 3 dose regimens of JS002 administered as multiple subcutaneous doses.
  Interventions: Biological: Biological：JS002
- Placebo (Placebo Comparator): Participants received matching placebo dose regimens by subcutaneous injection.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Biological：JS002 — Administered by subcutaneous injection
  Arms: JS002
Biological: Placebo — Administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
JS002 is a recombinant humanized anti-PCSK9 monoclonal antibody.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age ≥18 and ≤65 years old;
3. Body mass index (BMI) ≥18 and ≤ 30 kg/m2;
4. Subjects who are receiving statin therapy at the time of screening or who are eligible for statin therapy can receive a stable dose of statin therapy for more than 28 days before randomization and are willing to maintain stable statin therapy during the study;
5. Low-density lipoprotein cholesterol (LDL-C) level ≥2.6mmol/L for subjects who are receiving statin and/or other lipid-lowering therapy at the time of screening, or LDL-C≥ 4.1mmol/L for subjects who didn't receive any-lowering therapy at the time of screening, and LDL-C still ≥2.6mmol/L before randomization;
6. Fasting triglycerides ≤4.5 mmol/L;

Exclusion Criteria:

1. Diagnosis of homozygous familial hypercholesterolemia;
2. History of New York heart association (NYHA) defined Ⅱ - Ⅳ heart failure;
3. History of uncontrolled arrhythmiast;
4. History of myocardial infarction, history of PTCA or PCI or CABG, history of unstable angina befor 90 days of randomization;
5. History of stroke or TIA；
6. Uncontrolled hypertension with SBP≥160mmHg and/or DBP≥100mmHg
7. Type 1 diabetes, or type 2 diabetes that is or poorly controlled（HbA1c> 8.0%);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2020-05-03 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in low-density lipoprotein cholesterol (LDL-C) to week 12 | 12 weeks after the first dose

SECONDARY OUTCOMES:
Absolute value change from baseline in low-density lipoprotein cholesterol (LDL-C) | Twelve weeks after the last dose
Percent change from baseline in Total Cholesterol(TC、HDL-C、non-HDL-C、VLDL-C、Apo B、Apo A1、Lp(a) and TG ) | Twelve weeks after the last dose
Percentage change from baseline TC/HDL-C ratio | Twelve weeks after the last dose
Percent change from baseline in Apolipoprotein B (Apo B) | Twelve weeks after the last dose
Percent change from baseline in Apolipoprotein A-I (ApoA-I) | Twelve weeks after the last dose

OTHER OUTCOMES:
Number of subjects who develop detectable anti-drug antibodies (ADAs) | Twelve weeks after the last dose
Serum concentrations of JS002 | Twelve weeks after the last dose
Change from baseline in proprotein convertase total / free pcsk9 | Twelve weeks after the last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, China